CLINICAL TRIAL: NCT07361640
Title: DiaMester: E-health Lifestyle Program for Improved Self-management and Remission of Type 2 Diabetes - a Pilot RCT
Brief Title: DiaMester Pilot RCT: E-health Lifestyle Program for Type 2 Diabetes
Acronym: DiaMester
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Tromso (Other); Abel Technologies AS (Unknown); The Dam Foundation (Other); Diabetes Wellness Norway (Unknown); Norwegian Diabetes Association (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Anne-Marie Aas, Associate Professor and Clinical Dietitian, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 891668; SDAM_FOR555606 (Other Grant/Funding Number: The DAM foundation)
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; diabetes mellitus type 2; e-health; self-management; weight loss; low calorie diet; remission induction; total diet replacement; caloric restriction; diet therapy; health psychology; eating disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Loss; Feeding and Eating Disorders | interventions — Caloric Restriction

STUDY DESIGN:
Intervention Model Description: This registration covers a three-arm, parallel-group pilot RCT. Participants will be randomized in a 1:1:1 ratio to one of the two e-health lifestyle intervention arms or to the control group. The intervention and follow-up period is 1 year.
  The three arms include:
  1. e-health program with an LCD TDR of 750-900 kcal/day for a 3-month induction phase, aiming at 10-15% weight loss within 12 months,
  2. e-health program alone (without LCD) aiming at 10-15% weight loss within 12 months,
  3. control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): E-health program with LCD
  Interventions: Behavioral: e-health lifestyle program; Behavioral: Low calorie diet
- 2 (Experimental): E-health program without LCD
  Interventions: Behavioral: e-health lifestyle program
- 3 (No Intervention): Standard care, but with continuous glucose monitoring (CGM) for 10 days at baseline and 1 year.

INTERVENTIONS:
Behavioral: e-health lifestyle program — The e-health lifestyle program consists of three parts:
  1. an educational digital course module that can be tailored to the users' individual needs and preferences. This will include videos and interactive webinars accessible through the program, hosted by health specialists with users as guests.
  2. individual and group-based digital lifestyle coaching by trained health care personnel through secure video-conference and chat solutions.
  3. a mobile-phone-based self-management app. This app will offer the user relevant data and information from glucometer and smart watch according to the users' needs and preferences as well as easy ways for recording dietary intake, physical activity and other relevant parameters.
  Other Names: Lifestyle intervention; e-health based intervention; m-health intervention; digital behavioural intervention; weight loss intervention; total diet replacement low caloric diet
  Arms: 1; 2
Behavioral: Low calorie diet — Participants will use a low calorie diet (LCD) total diet replacement (TDR) for the first 3 months of the 1 year intervention period, before gradual reintroduction of food.
  Arms: 1

SUMMARY:
This registration covers a pilot for a 3-armed parallel-group randomized controlled trial (RCT) that will evaluate the efficacy of DiaMester, a Norwegian e-health programme designed to improve self-management and induce clinically meaningful weight loss, and thereby potential remission in adults with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The aim of this pilot RCT is to test the feasibility of the program and to investigate to what extent the program contributes to the intended improvement in lifestyle, self-management, metabolic risk factors and body weight. We also aim to investigate if participants in the e-health program achieve a clinically meaningful weight loss in each of the two intervention arms: one including a low-calorie diet (LCD) total diet replacement (TDR) induction phase and one without the use of a LCD.

The DiaMester app serves as a secure communication platform between each participant and an assigned health coach, who provides individually tailored advice on diet and physical activity and monitors progress towards agreed weight-loss targets. Six health coaches (clinical dietitians or diabetes nurses) will deliver the intervention, each having completed the same standardized training prior to study start.

Hypotheses:

Primary objective: To test whether participation in the DiaMester e-health program with an LCD induction phase results in greater weight loss compared to usual care after 12 months.

H1: The e-health + LCD group will achieve greater weight loss after 12 months than the control group

Secondary objectives:

A. To test whether participation in the DiaMester e-health program alone (without LCD) results in greater weight loss compared to usual care after 12 months.

H2: The e-health-only group will achieve greater weight loss than the control group after 12 months

B. Secondary outcomes include diet quality, lifestyle, physical activity, metabolic risk factors, and health related quality of life (HRQoL), self-management, eating disorder symptoms and diabetes distress. Both the LCD and no LCD intervention groups will be compared with the control group (usual care).

We hypothesize that compared to usual care, the e-health program supported lifestyle interventions will H3: Improve diet quality (in line with dietary recommendations), lifestyle index score and increase participants' physical activity H4: Improve the metabolic risk factors HbA1c, blood lipids, and blood pressure, H5: Reduce the use of blood glucose/lipid lowering drugs and/or blood pressure lowering drugs H5: Increase HRQoL and self-management and lower the level of diabetes distress.

H6: Not increase eating disorder symptoms

C: To examine possible mediating and moderating factors for the effect on body weight and metabolic risk factors H6: The intervention's effect on bodyweight is mediated by change in diet quality and physical activity H7: The intervention's effect on HbA1c, blood lipids and blood pressure is mediated by change in bodyweight, diet quality and physical activity H8: The effect of weight loss on HbA1c is moderated by diabetes duration, BMI and age

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Men and women aged ≥ 18 years
* Type 2 diabetes of duration 0-6 years (diagnosis based on 2 recorded diagnostic-level tests, HbA1c and/or blood glucose)
* HbA1c ≥ 48 mmol/mol at the last routine clinical check, within last 12 months if on diet alone
* HbA1c ≥ 43 mmol/mol if on treatment with oral hypoglycaemic agents or GLP-1 RA treatment
* Body Mass Index (BMI) >27 kg/m2
* Stable body weight during the last 6 months with or without the use of weight-reducing drugs
* Self-reported desire to lose weight
* Owns a smartphone

Exclusion criteria:

* Current insulin use
* > 5% weight change or started treatment with weight reducing drugs* within the last 6 months. *orlistat (Xenical), bupropion-naltrekson (Mysimba), fenteramin-topiramat (Qsimba), semaglutid (Wegovy, Ozempic), tirzepatid (Mounjaro), liraglutid (Saxenda, Victoza), dulaglutid (Truicity).
* Recent routine HbA1c ≥108 mmol/mol
* Recent eGFR <30 ml/min/1.73 m^2
* Known cancer
* Myocardial infarction within previous 6 months
* Severe heart failure defined as equivalent to the New York Heart Association grade 3 (NYHA)
* Pregnancy/considering pregnancy or exclusively breastfeeding
* Substance abuse (drugs, alcohol)
* Diagnosed eating disorders or suspected ED based on screening questionnaire
* Learning difficulties or unable to understand, speak and read Norwegian or English
* Patients who have required hospitalization for depression or are on antipsychotic drugs
* People currently participating in another clinical research trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline (weight loss) | Body weight will be assessed at baseline, 3 months, 6 months, 9 months and 12 months.
  Body weight (kg) will be measured by the participants' GPs. Change in body weight will be reported as percentage weight loss and will be analysed as a continuous variable.

SECONDARY OUTCOMES:
Change in HbA1c from baseline | HbA1c will be measured at baseline, 3 months, 6 months, 9 months and 12 months.
  HbA1c (mmol/mol) will be measured by the participants GPs and will be analysed as a continuous variable.
Change in blood lipids from baseline | Lipids will be measured at baseline, 6 months and 12 months
  Lipids (mmol/L) (total cholesterol, low density cholesterol, high density cholesterol, triglycerides, non-high density cholesterol) will be measured by the participants GPs and will be analysed as a continuous variable.
Change in blood pressure from baseline | Blood pressure will be measured at baseline, 3 months, 6 months, 9 months and 12 months.
  Change in blood pressure (mmHg) will be measured by the participants GPs and will be analysed as a continuous variable.
Change in blood glucose time in range from baseline | Participants' in the control group will wear a CGM for 10 days at baseline and 1 year, while participants' in the two intervention groups will wear a CGM for 40 days at baseline, 40 days at 6 months and 10 days at one year.
  Average blood glucose will be collected form continuous glucose monitors (CGM).
Change in average blood glucose baseline | Participants' in the control group will wear a CGM for 10 days at baseline and 1 year, while participants' in the two intervention groups will wear a CGM for 40 days at baseline, 40 days at 6 months and 10 days at one year.
  Average blood glucose will be collected form continuous glucose monitors (CGM).
Change in use of medications from baseline | Use of medications will be assessed at baseline, 3 months, 6 months, 9 months and 12 months.
  Type of blood glucose lowering drugs, lipid lowering drugs and blood pressure lowering drugs. We will report how many participants that are using zero, one and more than one glucose lowering drug, lipid lowering drug and blood pressure lowering drug. In addition, we will report the number of participants that are using GLP-1 analogues.
Change in diet quality from baseline | Diet quality will be assessed at baseline, 6 months and 1 year.
  Data on diet quality will be collected using 24 hour recall for 3 separate days at each time point. The Norwegian Diet Index (1) will be adapted to create a new index reflecting the Norwegian dietary guidelines for diabetes and the European recommendations for the dietary management of diabetes (The Diabetes and Nutrition Study Group of the EASD 2023). In addition, intake of nutrients and key food groups will be evaluated.
Change in physical activity from baseline | Physical activity will be assessed at baseline and 1 year follow up.
  Physical activity will be scored on the short form of the International physical activity questionnaire (IPAQ-SF) (2). For participants in the intervention groups physical activity (energy expenditure and steps) will be recorded with smart watches.
Change in health related quality (HRQoL) of life from baseline | Measured at baseline and 1 year follow-up
  HRQoL will be measured using the EQ-5D-5L (3).
Change in diabetes distress of life from baseline | Measured at baseline and 1 year follow-up
  Diabetes distress will be measured using the problem Areas in Diabetes Scale (PAID) (4) and/or the Diabetes Distress Scale (DDS) (5).
  Time frame: Measured at baseline and 1 year follow-up
Change in diabetes self-management from baseline | Measured at baseline and 1 year follow-up
  Diabetes self-management will be measured using the problem Diabetes Empowerment Scale-Short Form (DES-SF) (6).
Change in eating disorder symptoms from baseline | Measured at baseline and 1 year follow-up
  Eating disorder symptoms will be measured using the Eating Disorder Examination Questionnaire (EDE-Q) (7, 8). Individuals with a score indicating high likelihood of ED at baseline will undergo an interview evaluating diagnostic criteria.
Prevalence of likely eating disorder at baseline | Measured at baseline
  Eating disorder symptoms will be measured using the problem EDE-Q. Individuals with a score indicating high likelihood of ED at baseline will undergo an interview evaluating diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Aas, PhD, Principal Investigator — Oslo University Hospital and University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, as participants have not consented to data sharing beyond the purposes of the present study, and the data contain sensitive health information protected under GDPR.

REFERENCES:
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Polonsky WH, Anderson BJ, Lohrer PA, Welch G, Jacobson AM, Aponte JE, Schwartz CE. Assessment of diabetes-related distress. Diabetes Care. 1995 Jun;18(6):754-60. doi: 10.2337/diacare.18.6.754. PMID 7555499
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Henriksen HB, Berg HB, Andersen LF, Weedon-Fekjaer H, Blomhoff R. Development of the Norwegian diet index and the Norwegian lifestyle index and evaluation in a national survey. Food Nutr Res. 2023 Sep 29;67. doi: 10.29219/fnr.v67.9217. eCollection 2023. PMID 37808205